CLINICAL TRIAL: NCT04334070
Title: Novartis Multiple Patient Program for Lamprene® (Clofazimine) for the Treatment of Non-Tuberculous Mycobacterial (NTM) Infections
Brief Title: Lamprene Multiple Patient Program
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLAM320B2002M
Record Dates: First submitted 2020-04-02; First posted 2020-04-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Non-Tuberculous Mycobacterial (NTM) Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Lamprene®/Clofazimine — All participants will receive Lamprene/clofazimine 50 mg capsules. The recommended dose of clofazimine for this program is 100 mg once daily, administered orally, preferably with meals. Duration of treatment will be decided by the treating physician. When considering clofazimine for the treatment of NTM infection, clofazimine is to be administered as part of a multi-drug regimen.

SUMMARY:
Lamprene®/Clofazimine, is a product of the pharmaceutical company named Novartis Pharmaceuticals Corporation. Lamprene®/Clofazimine is approved by FDA (the U.S Food and Drug Administration) for the treatment of leprosy. It is no longer available through pharmacies in the US. It is being tested in non-Novartis clinical studies for drug resistant tuberculosis and non-tuberculous mycobacteria (NTM).

To be eligible for participation in this expanded access program, patients must have an NTM diagnosis. The treating physician has decided that this infection can be treated with Lamprene®/Clofazimine. This medicine is provided to the physician in an expanded access program. This means that this medicine is not registered for the treatment of NTM, but it can be used in special situations where there are no other possible treatments. For example, this may be because the patient has a type of Mycobacterial infection that is resistant or failed to respond optimally to other drugs, or because the patient has had side effects that prevent the use of other drugs. The physician must submit a patient registration form to initiate the patient approval process.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age or older
2. Written informed consent must be obtained before any project specific assessment is performed.
3. Patients previously diagnosed with NTM infection with local or disseminated infection(i.e. patients with any NTM species at any site of infection)
4. Patients who failed or are intolerant of prior therapies or who have baseline macrolide resistance or for whom an appropriate regimen cannot otherwise be devised
5. Male patients (including vasectomized patients) who agree to use a condom during intercourse while taking clofazimine treatment and for at least 4 months after stopping treatment with clofazimine
6. Female patients of child-bearing potential with negative pregnancy test before clofazimine treatment initiation and who confirm no intention to become pregnant during the treatment with clofazimine, by using highly effective methods of contraception (methods that result in less than 1% pregnancy rates) while taking clofazimine treatment and for at least 4 months after stopping treatment with clofazimine

Exclusion Criteria:

1. History of hypersensitivity to any drugs or metabolites of similar chemical classes as clofazimine
2. History or current diagnosis of clinically significant ECG abnormalities that pose a safety risk for the patient, such as clinically significant cardiac arrhythmias (e.g.,sustained ventricular tachycardia, second or third degree heart block without a pacemaker)
3. History or additional risk factors for Torsades de Pointes such as heart failure, clinically relevant hypokalemia, familial long QT syndrome or known family history of Torsades de Pointes
4. Confirmed demonstration of resting QTcF >500 msec at screening
5. Any condition (social, psychiatric, or medical) which in the opinion of the treating physician would make participation in this MPP unsafe
6. Unable to swallow capsules
7. HIV-infected patients with disseminated NTM infection
8. Life expectancy less than 6 months
9. Pregnant or nursing (lactating) females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult